CLINICAL TRIAL: NCT02385227
Title: A Proof-of-Concept Study to Characterize Biomarkers of Tobacco Exposure, Product Use, and Urge-to-Smoke Following Short-Term Exclusive and Dual Ad Lib Use of Electronic Cigarettes in a Controlled Clinical Setting
Brief Title: Characterization of Biomarkers of Tobacco Exposure, Urge-to-Smoke Following Exclusive and Dual Ad Lib Use of Electronic Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lorillard Tobacco Company (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DaVinci
Record Dates: First submitted 2015-02-06; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Cohort A1 (Experimental): Exclusive blu™ e-cigarette A1
  Interventions: Other: Exclusive blu™ e-cigarette A1
- Cohort A2 (Experimental): Exclusive blu™ e-cigarette A2
  Interventions: Other: Exclusive blu™ e-cigarette A2
- Cohort A3 (Experimental): Exclusive blu™ e-cigarette A3
  Interventions: Other: Exclusive blu™ e-cigarette A3
- Cohort B1 (Experimental): Dual blu™ e-cigarette and usual brand B1
  Interventions: Other: Dual blu™ e-cigarette and usual brand B1
- Cohort B2 (Experimental): Dual blu™ e-cigarette and usual brand B2
  Interventions: Other: Dual blu™ e-cigarette and usual brand B2
- Cohort B3 (Experimental): Dual blu™ e-cigarette and usual brand B3
  Interventions: Other: Dual blu™ e-cigarette and usual brand B3
- Cohort C (Experimental): Nicotine product cessation C
  Interventions: Other: Nicotine product cessation C

INTERVENTIONS:
Other: Exclusive blu™ e-cigarette A1 — Classic Tobacco rechargeable e cigarette
  Arms: Cohort A1
Other: Exclusive blu™ e-cigarette A2 — Magnificent Menthol rechargeable e cigarette
  Arms: Cohort A2
Other: Exclusive blu™ e-cigarette A3 — Cherry Crush rechargeable e cigarette
  Arms: Cohort A3
Other: Dual blu™ e-cigarette and usual brand B1 — Classic Tobacco rechargeable e cigarette and a usual brand combustible cigarette
  Arms: Cohort B1
Other: Dual blu™ e-cigarette and usual brand B2 — Magnificent Menthol rechargeable e cigarette and a usual brand combustible cigarette
  Arms: Cohort B2
Other: Dual blu™ e-cigarette and usual brand B3 — Cherry Crush rechargeable e cigarette and a usual brand combustible cigarette
  Arms: Cohort B3
Other: Nicotine product cessation C — Nicotine cessation
  Arms: Cohort C

SUMMARY:
This is a randomized, open-label, forced-switch, parallel, proof-of-concept study to assess exposure to biomarkers of tobacco exposure following short-term ad lib use of three blu e-cigarette products. The primary objectives of this study are to:

1. Compare changes in selected urine and blood biomarkers of tobacco exposure within cohorts following a 5-day forced-switch from usual brand conventional combustible cigarettes to exclusive use of blu e-cigarettes, dual use of blu e cigarettes and the subject's usual brand combustible cigarette, or smoking cessation.
2. Compare changes in selected urine and blood biomarkers of tobacco exposure among cohorts following a 5-day forced-switch from usual brand conventional combustible cigarettes to exclusive use of a blu e cigarette, dual use of a blu e-cigarette and the subject's usual brand combustible cigarette, or smoking cessation.

The secondary objectives of this study are to:

1. Compare changes in selected physiological endpoints affected by tobacco exposure within cohorts during a 5-day forced-switch from usual brand conventional combustible cigarettes to exclusive use of blu e cigarettes, dual use of blu e cigarettes and the subject's usual brand combustible cigarette, or smoking cessation.
2. Compare changes in selected physiological endpoints affected by tobacco exposure among cohorts following a forced-switch to exclusive use of a blu e cigarette, dual use of a blu e-cigarette and the subject's usual brand combustible cigarette, or smoking cessation.
3. Determine daily nicotine consumption from blu e-cigarettes following exclusive use of blu e cigarettes or dual use of blu e-cigarettes and the subject's usual brand combustible cigarette over a 5-day period.
4. Assess the effectiveness of exclusive use of blu e-cigarettes or dual use of blu e-cigarettes and the subject's usual brand combustible cigarette to reduce the urge to smoke.
5. Assess subject opinions of various characteristics of blu e-cigarettes.
6. Assess the safety and tolerability of short-term use of blu e-cigarettes.

DETAILED DESCRIPTION:
Subjects checked in to the clinic on Day -2 and continued to smoke their usual brand cigarette ad lib through the evening of Day -1 upon request to the clinic staff. Baseline assessments were made from the morning of Day -1 through the morning of Day 1 prior to the start of randomized product use. On the morning of Day 1, subjects were randomized into one of the study arms noted above and post-baseline assessments were made through the morning of Day 6.

With limited exceptions, all product use was ad lib from 07:30 to 23:00 on Days -2 to 5. Smoking of cigarettes and use of the e-cigarette products were limited to separate sections of the clinic to minimize the chance for illicit product use and cross-contamination. Subjects randomized to the cessation arm were housed in a separate section of the clinic after randomization.

From Day 1 to the end of the study all subjects randomized to an e-cigarette cohort were allowed to carry the assigned product with them throughout the day and use their product ad lib within identified sections of the clinic. Subjects randomized to the dual-use cohorts were allowed to smoke no more than 50% of the number of cigarettes per day reported at Screening. Cigarettes were were provided to the subjects upon request to the study staff.

Daily product use of blu e-cigarettes and usual brand cigarettes was assessed on Days -1 through Day 5. Each blu e-cigarette was weighed prior to dispensing and following the return of the product and the estimated amount of nicotine delivered from each blu e-cigarette will be calculated by multiplying the weight difference (mg) by 2.4%.

Urine biomarkers of exposure and effect were assessed from 24-hour urine collections from the morning of Day -1 to the morning of Day 1 and from the morning of Day 5 to the morning of Day 6. Urine biomarkers of exposure included NNAL, nicotine equivalents (nic + 5), 3-HPMA, CEMA, 1-OHP, NNN, MHBMA, and S-PMA. The urine biomarker of effect included F2-isoprostane (8-iso-PGF2 Type III). Biomarker concentrations were adjusted for urine creatinine concentrations.

Blood biomarkers of exposure included COHb, nicotine, cotinine, and trans-3'hydroxycotinine. Samples were collected on Days -1, 1, 3, and 5 in the morning prior to the start of product administration and in the evening.

Other physiologic endpoints included spirometry (FVC and FEV1, assessed in the afternoon on Day -1 and Day 5, exhaled CO and NO measurements (assessed in the afternoon on Days -1, 1, 3, and 5), and blood pressure and pulse rate (assessed on Days -1 through 5 in the morning prior to the start of product administration and evening).

Questionnaires administered included the Fagerström Test for Nicotine Dependence and the Brief Wisconsin Inventory of Smoking Dependence Motives (Day -1), smoking urge (Days -1 through 5 in the morning prior to the start of product administration and evening), and the Modified Cigarette Evaluation Scale (evening of Day 5, not administered to subjects in the cessation arm).

Safety evaluations included physical examinations, vital signs, ECGs, clinical laboratory assessments (clinical chemistry, hematology, urinalysis, and serology), urine drug and alcohol screens, urine cotinine and exhaled CO screens, and pregnancy tests (females only). Adverse events spontaneously reported by the subjects or observed by the Investigator or other study personnel were monitored from the time of Check-in until the End-of-Study (or Early Termination). Any concomitant medications taken from 30 days prior to Check-in through the End-of-Study (or Early Termination) were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and female smokers, 21 to 65 years of age, inclusive, at Screening.
2. Combustible cigarette smoker for at least 12 months prior to Check-in. Brief periods of non-smoking during the 90 to 14 days prior to Check-in (e.g., up to ~7 consecutive days due to illness, trying to quit, participation in a study where smoking was prohibited) will be permitted at the discretion of the Investigator.
3. Currently smokes an average of 10 or more king size (~83 - 85 mm) or 100s (~98 - 100 mm) manufactured combustible cigarettes per day (any brand style).
4. Consistent use of a single brand style for 14 days prior to Check-in.
5. Positive urine cotinine at Screening (≥ 500 ng/mL).
6. Exhaled CO > 12 ppm at Screening.
7. Female subjects of non-childbearing potential and of childbearing potential will be eligible. Examples of acceptable forms of contraception include, but are not limited to, the following.

   * Surgeries:Hysterectomy at least 6 months prior to product administration; Oophorectomy at least 6 months prior to product administration; Tubal ligation at least 6 months prior to product administration
   * Transcervical sterilization at least 6 months prior to product administration
   * Hormonal birth control at least 3 months prior to product administration
   * Non-hormonal intrauterine device at least 3 months prior to product administration
   * Double barrier methods (e.g., condom and spermicide) at least 14 days prior to product administration
   * Abstinence at least 14 days prior to product administration
   * Vasectomized partner is acceptable birth control for females provided the surgery was performed at least 6 months prior to product administration
   * Postmenopausal at least 1 year prior to product administration and confirmed by follicle stimulating hormone (FSH) test at Screening.
8. Understands the study procedures and provides voluntary consent to participate in the study documented on the signed ICF.
9. Willing to comply with the study requirements, including potential use of any study product or smoking cessation during the study.

Exclusion Criteria:

1. History or presence of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, pulmonary (especially bronchospastic diseases), immunologic, psychiatric, or cardiovascular disease, or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. Clinically significant abnormal findings on the physical examination, medical history, ECG, or clinical laboratory results at Screening or Check-in, in the opinion of the Investigator.
3. Positive test for HIV, HbsAg, or HCV.
4. An acute illness (e.g., upper respiratory infection, viral infection) requiring treatment within 2 weeks prior to Check-in.
5. Fever (>100.2F) at Screening or at Check-in.
6. Systolic blood pressure >150 mmHg, diastolic blood pressure >95 mmHg, or pulse rate >99 bpm at Screening.
7. BMI <18 kg/m2 or >40 kg/m2 at Screening.
8. Female subjects who are pregnant, lactating, or intend to become pregnant from Screening through completion of study.
9. Use of prescription anti-diabetic medication and/or insulin therapy within 12 months of Check-in.
10. Use of medications or foods known or are suspected to interact with cytochrome P450 2A6 (including, but not limited to, amiodarone, amlodipine, amobarbital, buprenorphine, clofibrate, clotrimazole, desipramine, disullfiram, entacapone, fenofibrate, isoniazid, grapefruit, ketoconazole, letrozole, methimazole, methoxsalen, metyrapone, miconazole, modafinil, orphenadrine, pentobarbital, phenobarbital, pilocarpine, primidone, propoxyphene, quinidine, rifampicin, rifampin, secobarbital, selegiline, sulconazole, tioconazole, tranylcypromine,) within 14 days or five half-lives of the drug, whichever is longer, prior to Check-in.
11. Use of inhalers to treat any medical condition within 3 months prior to Check-in and throughout the study.
12. Positive urine screen for alcohol or drugs of abuse at Screening or at Check-in.
13. History of drug or alcohol abuse within 24 months prior to Check-in.
14. Plasma donation within 7 days prior to Check-in.
15. Donation of blood or blood products, had significant blood loss, or received whole blood or a blood product transfusion within 56 days prior to Check-in.
16. Participation in a previous clinical study for an investigational drug, biologic, medical device, or tobacco product within 28 days prior to Check-in.
17. Use of tobacco or nicotine-containing products (e.g., roll-your-own cigarettes, bidis, snuff, snus, tablets, inhalers, pipes, cigars, chewing tobacco, nicotine replacement therapies [e.g., gum, patches, lozenges, nasal spray, or inhalers]) other than manufactured cigarettes or e-cigarettes within 28 days prior to Check-in.
18. Use of any prescription smoking cessation treatments, including, but not limited to, varenicline (Chantix) or buproprion (Zyban) within 3 months prior to Check-in.
19. Known hypersensitivity to the study products, glycerol, or propylene glycol.
20. Self-reported puffers (i.e., smokers who draw smoke from the cigarette into the mouth and throat but do not inhale).
21. Subject or a first-degree relative (i.e., parent, sibling, child) is a current or former employee of the tobacco industry or a named party or class representative in litigation with the tobacco industry.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Biomarkers of tobacco exposure as measured in urine | 5 days
  Excretion of each urine biomarker of exposure (NNAL, nicotine equivalents, 3-HPMA, HMPMA, CEMA, 1-OH pyrene, NNN, MHBMA, and S-PMA) will be assessed at baseline and following a 5-day forced switch to determine changes associated with product use or cessation, and differences between cohorts.
Biomarkers of tobacco effect as measured in urine | 5 days
  Excretion of F2-isoprostane (8-iso-PGF2 Type III) will be assessed at baseline and following a 5-day forced switch to determine changes associated with product use or cessation, and differences between cohorts.
Biomarkers of tobacco exposure as measured in blood | 5 days
  Exposure to each blood biomarker of exposure (COHb, nicotine, cotinine, and trans-3'hydroxycotinine) will be assessed at baseline and during a 5-day forced switch to determine changes associated with product use or cessation, and differences between cohorts.

SECONDARY OUTCOMES:
Daily product consumption as measured by e-cigarette and combustible cigarette use | 5 days
  Daily nicotine consumption from blu e-cigarettes and the number of cigarettes smoked per day will be assessed at baseline and during a 5-day forced switch to determine changes associated with product use and differences between cohorts.
Urge to smoke as measured by visual analog scale | 5 days
  The urge to smoke will be assessed at baseline and during a 5-day forced switch to determine the effectiveness of blu e-cigarettes to determine changes associated with product use or cessation, and differences between cohorts.
Physiologic effects as measured by spirometry | 5 days
  FVC and FEV1 will be assessed at baseline and during a 5-day forced switch to determine changes associated with product use or cessation, and differences between cohorts.
Physiologic effects as measured by exhaled breath | 5 days
  Exhaled CO and NO will be assessed at baseline and during a 5-day forced switch to determine changes associated with product use or cessation, and differences between cohorts.
Physiologic effects as measured by blood pressure and pulse rate | 5 days
  Sytolic and diastolic blood pressure and heart rate will be assessed at baseline and during a 5-day forced switch to determine changes associated with product use or cessation, and differences between cohorts.
Relationship between product use and biomarker exposure | 5 days
  The relationship between product use and exposure to the urine and blood biomarkers of tobacco exposure and effect will be assessed.
Subjective product assessments as measured by the modified cigarette evaluation scale | 5 days
  The Modified Cigarette Evaluation Scale will be administered to assess differences in subjective opinions of the blu e-cigarettes between cohorts.
Safety and tolerability as measured by number of subjects with adverse events or changes in health status | 5 days
  The safety and tolerability of blu e-cigarettes during a 5-day period of use will be assessed using physical examinations, vital signs, clinical laboratory assessments, and adverse event and concomitant medication monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Gartner, M.D., Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States

REFERENCES:
- [Derived] D'Ruiz CD, Graff DW, Robinson E. Reductions in biomarkers of exposure, impacts on smoking urge and assessment of product use and tolerability in adult smokers following partial or complete substitution of cigarettes with electronic cigarettes. BMC Public Health. 2016 Jul 11;16:543. doi: 10.1186/s12889-016-3236-1. PMID 27401980